CLINICAL TRIAL: NCT05499026
Title: Retrospective Cohort Study to Investigate the Safety and Efficacy of Chenodeoxycholic Acid (CDCA) in Patients Affected by Cerebrotendinous Xanthomatosis (CTX)
Brief Title: Safety and Efficacy of CDCA in CTX Chenodeoxycholic Acid (CDCA) in Patients Affected by Cerebrotendinous Xanthomatosis (CTX)
Status: Completed | Type: Observational
Sponsor: Leadiant Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CDCA-STUK-15-001
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Cerebrotendinous Xanthomatoses
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous | interventions — Chenodeoxycholic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chenodeoxycholic Acid — Bile acid

SUMMARY:
Retrospective study of CTX patients to investigate the safety and clinical efficacy of Chenodeoxycholic Acid

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of CTX Received treatment with CDCA Age between 2 and 75 years Having at least one cholestanol level and/or urinary bile alcohol level no more than 3 months prior to treatment with CDCA and one cholestanol level and/or urinary bile alcohol level post-treatment within 2 years from the beginning of therapy with CDCA

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: CTX patients
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2015-06-03 (Actual)

PRIMARY OUTCOMES:
Serum Cholestanol Levels | 34 years

IPD SHARING:
Plan to Share IPD: No